CLINICAL TRIAL: NCT03575156
Title: Microparticles's Role in the Pathophysiology of Systemic Lupus Erythematosus and Systemic Sclerosis
Acronym: MICROLUPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2017/54
Record Dates: First submitted 2018-06-07; First posted 2018-07-02 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Systemic Lupus Erythematosus; Systemic Scleroderma
Keywords: Systemic Lupus Erythematosus; Systemic Scleroderma; autoimmunity; microparticles; platelets
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic; Autoimmune Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic lupus erythematosus (SLE) (Experimental)
  Interventions: Biological: blood sample; Biological: urine sample
- systemic scleroderma (SSc) (Experimental)
  Interventions: Biological: blood sample; Biological: urine sample

INTERVENTIONS:
Biological: blood sample — 36 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation
Biological: urine sample — 6 ml

SUMMARY:
Our study aims at defining the role of circulating microparticles in the physiopathology of two rare auto-immune diseases: systemic lupus erythematosus (SLE) and systemic scleroderma (SSc). Microparticles might have an prognostic and diagnostic interest as well as potential for the discovery of new therapeutic strategies.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) and systemic scleroderma (SSc) are two rare and potentially life-threatening auto-immune systemic diseases. There is an urgent need to describe prognostic factors and to discover new therapeutic pathways. Microparticles (MPs) are small extracellular vesicles formed from activated cells including endothelial cells and platelets. Preliminary data from our lab indicate that these MPs might play a key role in SLE and SSc physiopathology. In fact, MPs from patients with SLE aggregates with T regulator lymphocytes (LTregs) and decrease their activity, thereby promoting auto-immunity. Some works also indicate that MPs might cargo DNA to the immune system, also promoting auto-immunity. The investigators hypothesized that MPs levels might be a prognostic factor in SLE and SSc and that studying the molecular mechanisms involved could provide new therapeutic targets.

Our study will recruit 100 patients with SLE or SSc followed in Bordeaux University Hospital. Among classical disease activity information, blood and urine samples will be collected at each visit to study circulating microparticles. Fundamental research will be realized on patients' sample to study molecular mechanisms involved.

Clinical and biological disease activity, treatment and outcomes will be studied in correlation with MPs to describe their potential prognostic role. Patients will be followed at regular intervals as their usual follow-up would request. No extra visit will be needed and blood samples will be drawn at the same times as those drawn for clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of systemic lupus erythematosus or systemic sclerosis;
* age ≥ 18 years;
* being affiliated to health insurance, willing to participate and to sign informed consent.

Exclusion Criteria:

* pregnant or breastfeeding women;
* patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Change in quantitative levels of circulating MPs between baseline and 12 months in the blood and urine samples of SLE and SSc patients | At baseline (Day 0) and 12 months from baseline

SECONDARY OUTCOMES:
Disease activity scores for SLE patients | At baseline (Day 0) and 12 months from baseline
  Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)
Disease activity scores for SSc patients | At baseline (Day 0) and 12 months from baseline
  Rodnan score
Quantification of P-selectin levels (soluble and on platelets) in the blood and urine samples of SLE and SSc patients | At baseline (Day 0) and 12 months from baseline
Quantification of FAS-ligand levels in the blood and urine samples of SLE and SSc | At baseline (Day 0) and 12 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christophe RICHEZ, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de rhumatologie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No